CLINICAL TRIAL: NCT00731939
Title: Titan® One Touch Release Inflatable Penile Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DK057CC
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Results first posted 2014-04-14 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-03

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Penile implant; Titan
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Titan® OTR IPP (Other): Subjects implanted with Titan® One Touch Release (OTR) Inflatable Penile Prosthesis (IPP)
  Interventions: Device: Inflatable Penile Prosthesis

INTERVENTIONS:
Device: Inflatable Penile Prosthesis — Hydraulic system designed to be surgically implanted into the penis for the management of erectile dysfunction.
  Other Names: Titan®; Titan® OTR

SUMMARY:
The purpose of this study is to assess the ease of deflation of the Titan® OTR pump.

ELIGIBILITY:
Inclusion Criteria:

* Participant has an estimated life expectancy of more than 5 years
* Participant has been diagnosed with erectile dysfunction (impotence)
* participant is willing to have the Titan OTR IPP implanted
* Participant is able and willing to complete all follow-up visits and procedures indicated in the protocol

Exclusion Criteria:

* Participant is unable or unwilling to sign the Informed Consent Form and /or comply with all follow-up requirements according to the study protocol
* Participant had a previous penile prosthesis or prior penile enlargement surgeries
* Participant has a compromised immune system, such as systemic lupus erythematosus, discoid lupus, or scleroderma
* Participant has had a myocardial infarction or coronary artery stent placement within 2 months prior to treatment
* Participant currently has uncontrolled or severe diabetes or other disease significantly reducing wound healing ability
* Participant does not have the manual dexterity or mental ability to operate the pump
* Participant has chordee or priapism
* Participant has penile sensory neuropathy
* Participant has serious bleeding disorder

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2007-11; Primary Completion 2009-10 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Brock, MD, Principal Investigator — St Joseph's Hospital; Ricardo Munarriz, MD, Principal Investigator — Boston Medical Center; Lawrence Levine, MD, Principal Investigator — Rush Presbyterian; Chad Ritenour, MD, Principal Investigator — Emory Healthcare; LeRoy Jones, MD, Principal Investigator — Urology San Antonio; William Bogache, MD, Principal Investigator — Carolina Urologic Research Center; Dana Ohl, MD, Principal Investigator — Michigan Urology Center; David Ralph, MD, Principal Investigator — University College London Hospital
Locations (8):
- United States (6):
  - Emory Healthcare, Altanta, Georgia
  - Rush Presbyterian, Chicago, Illinois
  - Boston Medical Center, Boston, Massachusetts
  - Michigan Urology Center, Ann Arbor, Michigan
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology San Antonio, San Antonio, Texas
- St Joseph's Hospital, London, Ontario, Canada
- University College London Hospital, London, UK, United Kingdom

REFERENCES:
- [Result] Ohl DA, Brock G, Ralph D, Bogache W, Jones L, Munarriz R, Levine L, Ritenour C. Prospective evaluation of patient satisfaction, and surgeon and patient trainer assessment of the Coloplast titan one touch release three-piece inflatable penile prosthesis. J Sex Med. 2012 Sep;9(9):2467-74. doi: 10.1111/j.1743-6109.2012.02819.x. Epub 2012 Jul 3. PMID 22759540

RESULTS

PARTICIPANT FLOW:
Groups:
- Titan® OTR IPP: Subjects implanted with Titan® One Touch Release (OTR) Inflatable Penile Prosthesis (IPP)
  Inflatable Penile Prosthesis : Hydraulic system designed to be surgically implanted into the penis for the management of erectile dysfunction.
Period: Overall Study
Arm/Group | Titan® OTR IPP
Started | 124
Completed | 90
Not Completed | 34
Not completed — Adverse Event | 6
Not completed — Lost to Follow-up | 15
Not completed — Not implanted with study device | 9
Not completed — Withdrawal by Subject | 2
Not completed — Did not meet enrollment criteria | 2

BASELINE CHARACTERISTICS:
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 76
  >=65 years | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 124
Region of Enrollment [Number; unit: participants]
  United States | 71
  Canada | 27
  United Kingdom | 26

OUTCOME MEASURES:

1. Primary Outcome: Assess the Ease of Deflation of the Titan® OTR Pump
Description: The study's primary endpoint was to demonstrate that at least 64% of subjects were mostly or completely satisfied with the ability to deflate the device at the 6-month follow-up. The study's primary objective was to assess the ease of deflation of the Titan® OTR pump via subject questionnaire at 6-month follow-up. Subjects were asked via questionnaire how satisfied they were with ease of deflation of their implant. Success criteria was a response of "satisfactory" or "somewhat satisfactory". Other possible responses were "neither satisfactory nor unsatisfactory", "somewhat unsatisfactory", and "very unsatisfactory".
Time Frame: 6 months
Measure: Number; unit: % of participants meeting success criter
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 96
% of participants meeting success criter | 70.8

2. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 1
Description: Subject Satisfaction - overall function
Time Frame: 3 months post-surgery
Measure: Number; unit: % satisfactory or somewhat satisfactory
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 94
% satisfactory or somewhat satisfactory | 72.4

3. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 1
Description: Subject Satisfaction - overall function
Time Frame: 6 months post-surgery
Measure: Number; unit: % satisfactory or somewhat satisfactory
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 96
% satisfactory or somewhat satisfactory | 90.6

4. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 1
Description: Subject Satisfaction - overall function
Time Frame: 12 months post-surgery
Measure: Number; unit: % satisfactory or somewhat satisfactory
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 90
% satisfactory or somewhat satisfactory | 90.0

5. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 2
Description: Subject Satisfaction - soft enough to conceal when deflated
Time Frame: 3 months post-surgery
Measure: Number; unit: % satisfactory or somewhat satisfactory
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 94
% satisfactory or somewhat satisfactory | 62.8

6. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 2
Description: Subject Satisfaction - soft enough to conceal when deflated
Time Frame: 6 months post-surgery
Measure: Number; unit: % satisfactory or somewhat satisfactory
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 96
% satisfactory or somewhat satisfactory | 76.0

7. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 2
Description: Subject Satisfaction - soft enough to conceal when deflated
Time Frame: 12 months post-surgery
Measure: Number; unit: % satisfactory or somewhat satisfactory
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 90
% satisfactory or somewhat satisfactory | 82.2

8. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 3
Description: Subject Satisfaction - ease of locating the deflation touch pads
Time Frame: 3 months post-surgery
Measure: Number; unit: % satisfactory or somewhat satisfactory
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 94
% satisfactory or somewhat satisfactory | 60.6

9. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 3
Description: Subject Satisfaction - ease of locating the deflation touch pads
Time Frame: 6 months post-surgery
Measure: Number; unit: % satisfactory or somewhat satisfactory
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 96
% satisfactory or somewhat satisfactory | 78.2

10. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 3
Description: Subject Satisfaction - ease of locating the deflation touch pads
Time Frame: 12 months post-surgery
Measure: Number; unit: % satisfactory or somewhat satisfactory
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 89
% satisfactory or somewhat satisfactory | 77.6

11. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 4
Description: Subject Satisfaction - ease of inflation
Time Frame: 3 months post-surgery
Measure: Number; unit: % satisfactory or somewhat satisfactory
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 94
% satisfactory or somewhat satisfactory | 68.1

12. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 4
Description: Subject Satisfaction - ease of inflation
Time Frame: 6 months post-surgery
Measure: Number; unit: % satisfactory or somewhat satisfactory
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 95
% satisfactory or somewhat satisfactory | 85.3

13. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 4
Description: Subject Satisfaction - ease of inflation
Time Frame: 12 months post-surgery
Measure: Number; unit: % satisfactory or somewhat satisfactory
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 88
% satisfactory or somewhat satisfactory | 86.4

14. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 5
Description: Subject Satisfaction - ease of deflation
Time Frame: 3 months post-surgery
Measure: Number; unit: % satisfactory or somewhat satisfactory
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 94
% satisfactory or somewhat satisfactory | 60.6

15. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 5
Description: Subject Satisfaction - ease of deflation
Time Frame: 6 months post-surgery
Measure: Number; unit: % satisfactory or somewhat satisfactory
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 96
% satisfactory or somewhat satisfactory | 70.8

16. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 5
Description: Subject Satisfaction - ease of deflation
Time Frame: 12 months post-surgery
Measure: Number; unit: % satisfactory or somewhat satisfactory
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 90
% satisfactory or somewhat satisfactory | 73.3

17. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 6
Description: Subject Satisfaction - hardness of erection when inflated
Time Frame: 3 months post-surgery
Measure: Number; unit: % satisfactory or somewhat satisfactory
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 94
% satisfactory or somewhat satisfactory | 82.0

18. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 6
Description: Subject Satisfaction - hardness of erection when inflated
Time Frame: 6 months post-surgery
Measure: Number; unit: % satisfactory or somewhat satisfactory
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 94
% satisfactory or somewhat satisfactory | 91.5

19. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 6
Description: Subject Satisfaction - hardness of erection when inflated
Time Frame: 12 months post-surgery
Measure: Number; unit: % satisfactory or somewhat satisfactory
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 89
% satisfactory or somewhat satisfactory | 93.2

20. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 7
Description: Subject Satisfaction - width when inflated
Time Frame: 3 months post-surgery
Measure: Number; unit: % satisfactory or somewhat satisfactory
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 94
% satisfactory or somewhat satisfactory | 77.6

21. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 7
Description: Subject Satisfaction - width when inflated
Time Frame: 6 months post-surgery
Measure: Number; unit: % satisfactory or somewhat satisfactory
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 94
% satisfactory or somewhat satisfactory | 86.1

22. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 7
Description: Subject Satisfaction - width when inflated
Time Frame: 12 months post-surgery
Measure: Number; unit: % satisfactory or somewhat satisfactory
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 89
% satisfactory or somewhat satisfactory | 79.8

23. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 8
Description: Subject Satisfaction - length when inflated
Time Frame: 3 months post-surgery
Measure: Number; unit: % satisfactory or somewhat satisfactory
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 94
% satisfactory or somewhat satisfactory | 54.3

24. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 8
Description: Subject Satisfaction - length when inflated
Time Frame: 6 months post-surgery
Measure: Number; unit: % satisfactory or somewhat satisfactory
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 95
% satisfactory or somewhat satisfactory | 61.1

25. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 8
Description: Subject Satisfaction - length when inflated
Time Frame: 12 months post-surgery
Measure: Number; unit: % satisfactory or somewhat satisfactory
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 90
% satisfactory or somewhat satisfactory | 68.9

26. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 9
Description: Subject Satisfaction - would you recommend this penile implant device to men with the same erectile difficulty that you had?
Time Frame: 3 months post-surgery
Measure: Number; unit: % responding "yes" and "probably"
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 94
% responding "yes" and "probably" | 79.8

27. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 9
Description: as for outcome 26
Time Frame: 6 months post-surgery
Measure: Number; unit: % responding "yes" and "probably"
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 96
% responding "yes" and "probably" | 86.5

28. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 9
Description: as for outcome 26
Time Frame: 12 months post-surgery
Measure: Number; unit: % responding "yes" and "probably"
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 90
% responding "yes" and "probably" | 87.8

29. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 10
Description: Subject Satisfaction - if you had the decision to make again, would you undergo this penile implant procedure again?
Time Frame: 3 months post-surgery
Measure: Number; unit: % responding "yes" and "probably"
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 94
% responding "yes" and "probably" | 72.4

30. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 10
Description: Subject Satisfaction - if you had the decision to make again, would you undergo this penile implant procedure again?
Time Frame: 6 months post-surgery
Measure: Number; unit: % responding "yes" and "probably"
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 96
% responding "yes" and "probably" | 83.3

31. Secondary Outcome: Evaluate User Acceptance of Titan® OTR - Question 10
Description: Subject Satisfaction - if you had the decision to make again, would you undergo this penile implant procedure again?
Time Frame: 12 months post-surgery
Measure: Number; unit: % responding "yes" and "probably"
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 90
% responding "yes" and "probably" | 86.7

32. Secondary Outcome: Assess the Ease of Implant of the Titan® OTR Question 1
Description: Titan OTR pre-implant product preparation was straightforward/simple?
Time Frame: At implant
Measure: Number; unit: percentage of responses
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 113
percentage of responses
  Completely disagree | 0.0
  Somewhat disagree | 0.0
  Neutral | 2.7
  Somewhat agree | 22.1
  Completely agree | 75.2

33. Secondary Outcome: Assess the Ease of Implant of the Titan® OTR - Question 2
Description: Titan OTR pre-implant product preparation was easier than your usual pump of choice?
Time Frame: At implant
Measure: Number; unit: percentage of responses
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 113
percentage of responses
  Completely disagree | 0.0
  Somewhat disagree | 0.0
  Neutral | 10.6
  Somewhat agree | 40.7
  Completely agree | 48.7

34. Secondary Outcome: Assess the Ease of Implant of the Titan® OTR - Question 3
Description: The subject was easily able to accommodate the OTR pump?
Time Frame: At implant
Measure: Number; unit: percentage of responses
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 113
percentage of responses
  Completely disagree | 0.0
  Somewhat disagree | 0.0
  Neutral | 2.7
  Somewhat agree | 20.4
  Completely agree | 77.0

35. Secondary Outcome: Assess the Ease of Training for Titan® OTR - Question 1
Description: It was easy for the subject to find the inflation bulb?
Time Frame: 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 108
percentage of participants
  Not at all | 0.0
  A little | 0.9
  Somewhat | 4.6
  Very | 13.9
  Extremely | 80.6

36. Secondary Outcome: Assess the Ease of Training for Titan® OTR - Question 2
Description: It was easy for the subject to find the deflation touch pads?
Time Frame: 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 108
percentage of participants
  Not at all | 1.9
  A little | 3.7
  Somewhat | 9.3
  Very | 26.9
  Extremely | 58.3

37. Secondary Outcome: Assess the Ease of Training for Titan® OTR - Question 3
Description: It was easy for the subject to inflate the device?
Time Frame: 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 108
percentage of participants
  Not at all | 1.9
  A little | 0.9
  Somewhat | 4.6
  Very | 17.6
  Extremely | 75.0

38. Secondary Outcome: Assess the Ease of Training for Titan® OTR - Question 4
Description: It was easy for the subject to compress the deflation touch pads?
Time Frame: 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 108
percentage of participants
  Not at all | 2.8
  A little | 1.9
  Somewhat | 10.2
  Very | 25.9
  Extremely | 59.3

39. Secondary Outcome: Assess the Ease of Training for Titan® OTR - Question 5
Description: Subject training with OTR pump was easier than with previous pump?
Time Frame: 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 108
percentage of participants
  Not at all | 1.9
  A little | 1.9
  Somewhat | 16.7
  Very | 16.7
  Extremely | 63.0

40. Secondary Outcome: Assess the Ease of Training for Titan® OTR - Question 6
Description: The OTR pump was easy to use at 1st cycling?
Time Frame: 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 108
percentage of participants
  Not at all | 1.9
  A little | 5.6
  Somewhat | 8.3
  Very | 21.3
  Extremely | 63.0

41. Secondary Outcome: Assess the Ease of Training for Titan® OTR - Question 7
Description: The subject likes the OTR pump?
Time Frame: 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 108
percentage of participants
  Not at all | 0.9
  A little | 3.7
  Somewhat | 13.0
  Very | 20.4
  Extremely | 62.0

42. Secondary Outcome: Assess the Ease of Training for Titan® OTR - Question 8
Description: How easy was it for the subject to learn?
Time Frame: 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 107
percentage of participants
  Not at all | 2.8
  A little | 8.4
  Somewhat | 7.5
  Very | 29.9
  Extremely | 51.4

43. Secondary Outcome: Assess the Ease of Training for Titan® OTR - Question 9
Description: How likely the subject will need continued training or retraining?
Time Frame: 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 107
percentage of participants
  Not at all | 5.6
  A little | 10.3
  Somewhat | 11.2
  Very | 25.2
  Extremely | 47.7

44. Secondary Outcome: Assess Partner Satisfaction (Where Applicable)
Description: The Partner Treatment Satisfaction Scale (TSS) was used. The TSS provides scores ranging from 0 to 100 in 5 domains of Ease of erection, Erectile function, Pleasure from sexual activity, Satisfaction with orgasm and Confidence to complete sexual activity with higher scores indicative of worse symptoms. Available data is summarized for each domain at each visit along with change from baseline.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 59
units on a scale
  Ease of erection | 22.9 (28.3)
  Erectile function | 18.1 (23.9)
  Pleasure from sexual activity | 35.6 (29.8)
  Satisfaction with orgasm | 35.2 (33.2)
  Confidence to complete sexual activity | 23.2 (27.0)

45. Secondary Outcome: Assess Partner Satisfaction (Where Applicable)
Description: as for outcome 44
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Titan® OTR IPP
Number analyzed (Participants) | 39
units on a scale
  Ease of erection | 67.8 (31.3)
  Erectile function | 74.8 (20.4)
  Pleasure from sexual activity | 64.7 (24.8)
  Satisfaction with orgasm | 62.2 (29.2)
  Confidence to complete sexual activity | 71.2 (28.4)

ADVERSE EVENTS:
Time Frame: 12 months
Description: The analysis is based on the per protocol population (n=113). Of 124 consented subjects, nine (9) subjects did not meet inclusion/exclusion criteria and were not implanted with the study device. Two (2) subjects did not meet enrollment criteria and these two subjects were not followed for safety or efficacy.
Arm/Group | Titan® OTR IPP
Serious Adverse Events (participants affected / at risk) | 10/113
Other Adverse Events (participants affected / at risk) | 14/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Titan® OTR IPP (N=113)
Infection (Surgical and medical procedures) | 4 (4)
Hematoma (Surgical and medical procedures) | 2 (2)
Device malfunction (Surgical and medical procedures) | 2 (2)
Chronic pain (Surgical and medical procedures) | 1 (1)
Cylinder extrusion (Surgical and medical procedures) | 1 (1)
Scrotal abscess (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Titan® OTR IPP (N=113)
Auto inflation (Surgical and medical procedures) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No